CLINICAL TRIAL: NCT01163968
Title: Maximizing Outcomes Needed After Percutaneous Coronary Intervention (PCI) Using Weight Management (MOMENTUM)
Acronym: MOMENTUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0177-09-FB; 1P20NR011404-01 (NIH)
Record Dates: First submitted 2010-07-06; First posted 2010-07-16 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: Weight reduction; Cardiac revascularization; Percutaneous Coronary Intervention; Cardiac Rehabilitation; Rural
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Magnesium Salicylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight reduction program (Experimental): MOMENTUM intervention
  Interventions: Behavioral: MOMENTUM

INTERVENTIONS:
Behavioral: MOMENTUM — The Maximizing Outcomes Needed After Percutaneous Coronary Intervention (PCI) Using Weight Management (MOMENTUM) intervention is comprised of 6 modules, totaling 52 daily sessions promoting weight reduction, and 4 coaching sessions over the duration of the 12 week MOMENTUM intervention. The MOMENTUM intervention will be delivered using telehealth methods (Viterion telehealth device will be used to deliver the module content and coaching sessions). The intervention was purposively designed to overcome access barriers by using delivery modes accessible to patients in rural settings, in their home and at times convenient to their schedule.

SUMMARY:
The purpose of this study is to examine the use of a home-based program to improve weight reduction after percutaneous coronary intervention (PCI) (either a cardiac stent or angioplasty procedure).

DETAILED DESCRIPTION:
Obesity is an independent risk factor for coronary disease and is prevalent among patients who undergo percutaneous coronary intervention (PCI). The significance of cardiac disease is often underestimated by patients who undergo PCI, and therefore they are more reticent in modifying their cardiac risk factors such as obesity following PCI. This issue is particularly problematic for rural populations, given that weight reduction specific programs are often not available in rural communities. The overall goal of this pilot study is to evaluate a 12 week cognitive behavioral intervention for weight reduction of overweight or obese PCI patients who participate in a rural cardiac rehabilitation (CR) program. The Maximizing Outcomes Needed After Percutaneous Coronary Intervention (PCI) Using Weight Management (MOMENTUM) intervention is comprised of 6 modules, totaling 52 daily sessions promoting weight reduction, and 4 coaching sessions over the duration of the 12 week MOMENTUM intervention. The MOMENTUM intervention will be delivered using telehealth methods (Viterion telehealth device will be used to deliver the module content and the telephone to deliver the coaching sessions). The intervention was purposively designed to overcome access barriers by using delivery modes accessible to patients in rural settings, in their home and at times convenient to their schedule. A randomized, 2-group, repeated measures experimental design will be used. Subjects who have had a PCI, are overweight or obese and enroll in a rural cardiac rehabilitation program will be randomized to either the MOMENTUM group (n=25) and or control group (usual care)(n=25). The primary aim of the study is to compare the differences between the groups on weight reduction (primary outcome), diet behavior and physical activity (secondary outcomes) over time (baseline, 16 weeks, 6 and 9 months after PCI). The second aim of the study is to to evaluate the feasibility of implementing the MOMENTUM intervention for a larger randomized controlled trial. The innovation in this pilot study is the use of technology to deliver a comprehensive cognitive-behavioral weight reduction program to those cardiac patients in rural communities who otherwise might not have access to specific weight reduction programs to improve their cardiac risk profile after an acute cardiac event, such as a PCI.

ELIGIBILITY:
Inclusion Criteria:

* The sample for the proposed study will be 50 overweight or obese adults who have had a PCI who meet the following criteria:

  * planning to participate in cardiac rehabilitation at rural study sites in Saline and Seward counties of Nebraska
  * enrolled within 5 days of PCI procedure
  * oriented to person, place, and time
  * not visually impaired and able to hear
  * have telephone service
  * cardiologist's approval to participate in this study.

Exclusion Criteria:

* Mental status impairment as determined by a score of > 8 on the Short-Portable Mental Status Questionnaire (SPMSQ)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2013-03-04 (Actual); Study Completion 2013-03-04 (Actual)

PRIMARY OUTCOMES:
Weight reduction | 16 weeks after PCI
  Body Weight
Weight reduction | 6 months after PCI
  Body Weight
Weight reduction | 9 months after PCI
  Body Weight

SECONDARY OUTCOMES:
Diet behavior | 16 weeks after PCI
  Heart Healthy Eating Self-Efficacy Scale
Physical Activity behavior | 16 weeks after PCI
  Actigraph: mean levels of moderate activity
Abdominal fat content percent (%) change | 16 weeks after PCI
  Waist Circumference
Diet behavior | 6 months after PCI
  Heart Healthy Eating Self-Efficacy Scale
Diet behavior | 9 months after PCI
  Heart Healthy Eating Self-Efficacy Scale
Physical Activity behavior | 6 months after PCI
  Actigraph: mean levels of moderate activity
Physical Activity behavior | 9 months after PCI
  Actigraph: mean levels of moderate activity
Abdominal fat content percent (%) change | 6 months after PCI
  Waist Circumference
Abdominal fat content percent (%) change | 9 months after PCI
  Waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Barnason, PhD, Principal Investigator — University of Nebraska
Locations (1):
- BryanLGH Medical Center, Lincoln, Nebraska, United States